CLINICAL TRIAL: NCT05471648
Title: Phase 1, Double-Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Trial of EirGenix' Pertuzumab and Perjeta® (Pertuzumab) Sourced From US and EU Administered to Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing EG1206A and Perjeta (Pertzumab) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EirGenix, Inc. (Industry)
Collaborators: Sacura GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGC101; 2021-006769-40 (EudraCT Number)
Record Dates: First submitted 2022-07-08; First posted 2022-07-25 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: HER2 positive; early stage breast cancer; metastatic breast cancer; combination therapy; inhibiting MAP Kinase; P13K/Akt
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; pertuzumab

STUDY DESIGN:
Intervention Model Description: Phase 1, Double-Blind, Randomized, Parallel-Group, Single-Dose, 3-Arm, Comparative Pharmacokinetic Trial of EirGenix' Pertuzumab and Perjeta® (Pertuzumab) sourced from US and EU Administered to Healthy Male Volunteers
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 420 mg EirGenix Pertuzumab (Experimental): EirGenix Pertuzumab given intravenous with an infusion bag as a single dose of 420 mg over 60min.
  Interventions: Drug: 420 mg EG1206A EirGenix Pertuzumab in 14 mL Injection
- 420 mg Pertuzumab Perjeta EU Origin (Active Comparator): EU Pertuzumab given intravenous with an infusion bag as a single dose of 420 mg over 60min.
  Interventions: Drug: Perjeta (EU origin) 420 mg in 14 mL Injection
- 420 mg Pertuzumab Perjeta US Origin (Active Comparator): US Pertuzumab given intravenous with an infusion bag as a single dose of 420 mg over 60min.
  Interventions: Drug: Perjeta (US origin) 420 mg in 14 mL Injection

INTERVENTIONS:
Drug: 420 mg EG1206A EirGenix Pertuzumab in 14 mL Injection — Healthy volunteers receive pertuzumab (EG1206A, 420 mg, single dose)
  Other Names: Pertuzumab
  Arms: 420 mg EirGenix Pertuzumab
Drug: Perjeta (EU origin) 420 mg in 14 mL Injection — Healthy volunteers receive pertuzumab (Perjeta (EU origin) 420 mg, single dose)
  Other Names: Pertuzumab
  Arms: 420 mg Pertuzumab Perjeta EU Origin
Drug: Perjeta (US origin) 420 mg in 14 mL Injection — Healthy volunteers receive pertuzumab (Perjeta (US origin), 420 mg, single dose)
  Other Names: Pertuzumab
  Arms: 420 mg Pertuzumab Perjeta US Origin

SUMMARY:
This trial is a single-center, single-dose, double-blind, parallel-group, randomized, 3-arm PK trial in healthy male volunteers comparing a biosimilar pertuzumab (EG1206A) to a single intravenous (i.v.) infusion to both European Union (EU) and United States of America (US) reference products.

DETAILED DESCRIPTION:
This trial is part of a clinical development program developing a biosimilar pertuzumab, comparing the PK, safety and tolerability and immunogenicity of pertuzumab after a single intravenous (i.v.) infusion.

It assess the bioequivalence, PK characteristics, safety and tolerability as well as the immunogenicity of a test preparation containing 420 mg pertuzumab (EG1206A EirGenix Pertuzumab) as compared to marketed reference (EU and US) after a single dose i.v. infusion over 60 minutes in fasted state.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 55 years
* overtly healthy as determined by medical evaluation
* Body weight of at least 50 kg and not higher than 105 kg at screening
* BMI above/equal to 18.0 and below/equal to 30.0 kg/m2 at screening
* Male
* Agrees to the following during the treatment period and until 3 months after administration:
* Be and remain abstinent from heterosexual intercourse OR agree to use a male condom and female partners of childbearing potential must use an additional highly effective contraceptive method
* Abstain from donating sperm.
* Signed informed consent
* Valid COVID-19 immunization status as per current regulations

Exclusion Criteria:

* History or evidence of any clinically relevant disease, as judged by the investigator
* Any medical disorder, condition, or history of such that would impair the participant's ability to participate or complete this trial in the opinion of the investigator
* Pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination, and effects of the IMP will not be normal
* Known or suspected hypersensitivity to the IMPs (active substances, or excipients of the preparations)
* Known severe allergies e.g., allergies to more than 3 allergens
* Relevant diseases within the last 4 weeks before IMP administration
* Febrile illness within 2 weeks before IMP administration.
* History of known or suspected malignant tumors
* Known or suspected disorder of the liver
* Use of systemic/topical medicines/substances which oppose the trial objectives, or which might influence them within 4 weeks before IMP administration
* Regular use of therapeutic or recreational drugs or supplements
* Use of any herbal products or St. John's wort from 4 weeks before IMP administration
* Prior treatment with pertuzumab
* Smoking
* History of alcohol or drug abuse
* Regular daily consumption of more than 500 mL of usual beer or the equivalent quantity of approximately 20 g of alcohol in another form
* Intake of alcohol containing food and beverages from 48 h prior to admission to the ward
* Regular daily consumption of more than 1 L of methylxanthine-containing beverages
* Excluded physical therapies that might alter the PK or safety results of the trial from 7 days before IMP administration until follow-up
* Strenuous physical exercise or sauna visit with 72 h before admission to the ward
* Donation of more than 100 mL of whole blood or plasma within 4 weeks or approximately 500 mL whole blood within 3 months before IMP administration
* Plasmapheresis within 3 months before IMP administration
* Previous or concomitant participation in another clinical trial with IMP(s)
* Clinically relevant findings in the ECG
* LVEF below 55%
* Systolic blood pressure below 100 mmHg or above 140 mmHg
* Diastolic blood pressure below 50 mmHg or above 90 mmHg
* Heart rate below 50 beats/ min or above 90 beats/min
* Clinically relevant findings in the physical examination that may affect the objectives of the trial, or the safety of the participant
* Poor venous access
* Clinically relevant deviations of the screened safety laboratory parameters
* Alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, gamma glutamyl transpeptidase, or total bilirubin above 1.2 upper limit of normal
* Thyroid disorders as evidenced by assessment of thyroid stimulating hormone (TSH) level outside the normal reference range
* Positive results for hepatitis B virus surface antigen, hepatitis C virus antibodies, human immune deficiency virus antibodies, and human immune deficiency virus antigen
* Positive urine drug test
* Positive alcohol test
* Positive cotinine test
* Any criteria which, in the opinion of the investigator, preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety
* Close affiliation with the investigational site
* Vulnerable participants who are e.g., institutionalized due to regulatory or juridical order dependent on sponsor, site, or investigator or not able to consent, respectively.
* History of COVID-19 within 2 months prior to screening
* Long COVID-19 syndrome or other clinically relevant COVID-19 related symptoms or sequelae
* Positive SARS-CoV-2 viral ribonucleic acid (RNA) test at admission
* No SARS-CoV-2 vaccinations should be booked within 14 days before IMP administration and until last trial visit.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 135 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
AUC0-inf of pertuzumab | Pre-dose to day 91, 21 timepoints
  Area under the plasma concentration-time curve, from time 0 h extrapolated to infinity

SECONDARY OUTCOMES:
Cmax | Pre-dose to day 91, 21 timepoints
  Peak plasma concentration of a pertuzumab after administration
tmax | Pre-dose to day 91, 21 timepoints
  Time to reach peak plasma concentration of pertuzumab after administration
t1/2 | Pre-dose to day 91, 21 timepoints
  Terminal elimination half-life
Drug clearance (CL) | Pre-dose to day 91, 21 timepoints
  Total clearance
Volume of distribution (Vd) | Pre-dose to day 91, 21 timepoints
  The apparent volume in which pertuzumab is distributed
AUC0-last of pertuzumab | Pre-dose to day 91, 21 timepoints
  Area under the plasma concentration-time curve, from time 0 h to last measured timepoint
Frequency of treatment-emergent adverse events (AEs) | Day 1 to day 91
Immunogenicity: Anti-drug antibodies (ADA) and neutralizing antibodies (NAb) | Pre-dose to day 91, 7 timepoints
  Analysis of anti-drug antibodies (ADA) and neutralizing antibodies (NAb; only assessed following confirmed positive ADA results)

OTHER OUTCOMES:
Local tolerability at infusion site | Day 1 to day 15, 14 timepoints
  Assessment at the injection site by visual inspection of local reactions at and around the injection site
Vital sign - blood pressure | Day 1 to day 91, 8 timepoints
  Blood pressure (systolic and diastolic) will be measured after the participant had rested at least 5 min rest in supine position
Vital sign - pulse rate | Day 1 to day 91, 8 timepoints
  Pulse rate will be measured after the participant had rested at least 5 min rest in supine position
Physical examination | Day -1 to day 91, 5 timepoints
  Physical examination (by means of inspection, palpation, auscultation) includes general condition/psyche, skin, lymph nodes, head (including eyes, ears, mouth), thyroid gland, and throat, lungs, heart, abdomen, musculoskeletal system, neurological system, and vascular system.
Electrocardiogram (ECG) measurements | Day 1 to day 91, 7 timepoints
  A standard 12-lead ECG will be recorded after at least 5 min rest in supine position calculating heart rate (HR), PR/PQ interval, QRS interval, QT interval (uncorrected), QT interval according to Bazett's formula (QTcB)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Berse, Dr. med., Principal Investigator — CRS Clinical Research Services Berlin GmbH
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No